CLINICAL TRIAL: NCT02180776
Title: A Randomized Crossover Pilot Study To Determine Clinical Effectiveness and Patient Wellness of Inelastic Lumbosacral Orthoses Versus Standard Medical Treatment in Patients With Back Pain AssociatEd With Kyphosis (The ARISE Study)
Brief Title: Effectiveness of Inelastic LSO Versus Standard Medical Treatment for Back Pain Associated With Kyphosis
Acronym: ARISE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aspen Medical Products (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CPR-ORTHO01-2012
Record Dates: First submitted 2014-01-23; First posted 2014-07-03 (Estimated); Last update posted 2014-07-03 (Estimated); Status verified 2014-07

CONDITIONS: Kyphosis; Back Pain
MeSH Terms: conditions — Kyphosis; Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Active Comparator): Patients assigned to group A wore the Summit 456 TLSO (intervention) for four weeks in phase 1 of the study, followed by four weeks of observation (control) in phase 2.
  Interventions: Other: Summit 456 TLSO
- Group B (Placebo Comparator): Patients assigned to group B started four weeks of observation (control) in phase 1, followed by four weeks of summit 456 TLSO (intervention) in phase 2 of the study.
  Interventions: Other: Summit 456 TLSO

INTERVENTIONS:
Other: Summit 456 TLSO — Thoracolumbarsacral orthosis

SUMMARY:
The objective of this study is to evaluate clinical effectiveness and the effect on quality of life of an inelastic thoracolumbarasacral orthosis in male and female hyperkyphotic patients with moderate to severe back pain disability and to demonstrate the safety of the intervention through detailed reporting and analysis of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Patients with moderate to complete disability (crippled) as defined by a score of 21% to 80% on the baseline evaluation of the Oswestry Back Pain Disability Questionnaire;
* Patients diagnosed with kyphosis and have a Cobb angle of at least 55 degrees;
* Willing and able to comply with the study procedures and provide written informed consent to participate in the study.

Exclusion Criteria:

* Patients under the age of 19;
* Pregnant patients or patients who are considering future pregnancies;
* Patients who were participating in any other investigational device or drug study or whose participation in a previous investigational study within 30 days of study entry may, in the opinion of the clinical investigator, impact analysis of this orthotic;
* Patients who, in the clinical judgment of the investigator, are not suitable for this study; Patients who, in the investigators opinion, are mentally or legally incapacitated preventing informed consent or unable to read or understand written material;
* Patients who are unable or unwilling to return to the study center for follow-up visits.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2012-06; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Mean difference in the Oswestry Disability Index Scores of the intervention versus control groups | 4 weeks

SECONDARY OUTCOMES:
Measured amount of opioid medication consumed in the intervention group versus control group | Baseline and weeks 2,3,4,8,12,16,20 and 24

OTHER OUTCOMES:
ODI scores between the intervention group versus control group | Weeks 8, 12, 16, 20 and 24
SF-26v2 Survey scores in the intervention versus the control group | Baseline and weeks 4, 8, 12 and 24.
Cost and return on investment of the LSO intervention | 24 weeks
Number of adverse events associated with the LSO intervention | Baseline and weeks 2, 3, 4, 8, 12, 16, 20 and 24

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J Schaffer, MD, Principal Investigator — Southeastern Integrated Medical